CLINICAL TRIAL: NCT01971567
Title: High-resolution, Relational, Resonance-based, Electroencephalic Mirroring (HIRREM) to Relieve Insomnia: A Randomized, Placebo-Controlled Clinical Trial
Brief Title: High-resolution, Relational, Resonance-based, Electroencephalic Mirroring (HIRREM) to Relieve Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00024763
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Insomnia
Keywords: Insomnia; Electroencephalic; Biofeedback; Neural oscillations; Auto calibration; Relaxation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- HIRREM (Active Comparator): High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM) is a novel, noninvasive, electroencephalic-based feedback technology to facilitate relaxation and auto-calibration of neural oscillations by using auditory tones to reflect brain frequencies in near real time.
  Interventions: Device: HIRREM
- Placebo (Placebo Comparator): Subjects in this arm will receive a sham-HIRREM placebo, for which the scalp sensors have no active recording capability, and for which the auditory tonal feedback is randomly generated rather than based on current brain frequencies and amplitudes.
  Interventions: Device: HIRREM

INTERVENTIONS:
Device: HIRREM
  Other Names: High-resolution, relational, resonance-based, electroencephalic mirroring; Brainwave Optimization

SUMMARY:
The purpose of this study is to determine whether the addition of High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM) to usual care will improve insomnia symptoms based on changes in the Insomnia Severity Index at two months following completion of the intervention, compared to placebo plus usual care.

DETAILED DESCRIPTION:
Insomnia is the most prevalent sleep disorder and is associated with significant psychosocial and somatic pathology. Effective noninvasive interventions for insomnia are lacking. High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM), is a noninvasive, brain feedback technology to facilitate relaxation and auto-calibration of neural oscillations by using auditory tones to reflect brain frequencies in near real time. An open label, randomized, crossover pilot trial showed that HIRREM was safe and effective, with significant benefits for individuals with moderate to severe insomnia, based on differential change with symptoms of insomnia (Insomnia Severity Index, ISI). This study will extend those results in a larger cohort using a single blind, placebo controlled study design.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe clinical insomnia (Insomnia Severity Index score of 15 or higher)

Exclusion Criteria:

* Unable, unwilling, or incompetent to provide informed consent
* Physically unable to come to the study visits
* Known obstructive sleep apnea
* Diagnosed periodic limb movement disorder or known restless legs syndrome
* Known seizure disorder
* Known urinary problem (i.e. benign prostatic hypertrophy) which is the likely cause of the sleep disturbance
* Severe hearing impairment
* Known, or suspected diagnosis of post-traumatic stress disorder (PTSD)
* Known, relevant traumatic brain injury (TBI)
* Ongoing need for treatment with opiate, benzodiazepine, or anti-psychotic medications, anti-depressant medications such as SSRI, SNRI, or tricyclics, and sleep medications such as zolpidem or eszopiclone
* Anticipated and ongoing use of recreational drugs or alcohol
* Lack of internet or smart phone access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2016-12-12 (Actual); Study Completion 2017-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles H. Tegeler, MD, Principal Investigator — Department of Neurology, Wake Forest School of Medicine
Locations (1):
- Department of Neurology, Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Gerdes L, Gerdes P, Lee SW, H Tegeler C. HIRREM: a noninvasive, allostatic methodology for relaxation and auto-calibration of neural oscillations. Brain Behav. 2013 Mar;3(2):193-205. doi: 10.1002/brb3.116. Epub 2013 Jan 14. PMID 23532171
- [Background] Tegeler CH, Kumar SR, Conklin D, Lee SW, Gerdes L, Turner DP, Tegeler CL, C Fidali B, Houle TT. Open label, randomized, crossover pilot trial of high-resolution, relational, resonance-based, electroencephalic mirroring to relieve insomnia. Brain Behav. 2012 Nov;2(6):814-24. doi: 10.1002/brb3.101. Epub 2012 Oct 28. PMID 23170244
- [Derived] Tegeler CL, Shaltout HA, Lee SW, Simpson SL, Gerdes L, Tegeler CH. High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM) improves symptoms and autonomic function for insomnia: A randomized, placebo-controlled clinical trial. Brain Behav. 2020 Nov;10(11):e01826. doi: 10.1002/brb3.1826. Epub 2020 Sep 17. PMID 32940419

RESULTS

PARTICIPANT FLOW:
Groups:
- HIRREM: High-resolution, relational, resonance-based, electroencephalic mirroring (HIRREM) is a novel, noninvasive, electroencephalic-based feedback technology to facilitate relaxation and auto-calibration of neural oscillations by using auditory tones to reflect brain frequencies in near real time.
  HIRREM
- Placebo: Subjects in this arm will receive a sham-HIRREM placebo, for which the scalp sensors have no active recording capability, and for which the auditory tonal feedback is randomly generated rather than based on current brain frequencies and amplitudes.
  HIRREM
Period: Overall Study
Arm/Group | HIRREM | Placebo
Started | 56 | 51
Completed | 52 | 49
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIRREM | Placebo | Total
Number analyzed (Participants) | 56 | 51 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (15.1) | 54.7 (14.8) | 53.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 32 | 73
  Male | 15 | 19 | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White | 46 | 43 | 89
  Ethnicity: Other | 10 | 8 | 18
Duration with Sleep Trouble [Mean (Standard Deviation); unit: years] | 11.1 (12.1) | 12.2 (11.3) | 11.7 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Insomnia Severity Index (ISI)
Description: The ISI is a 7 question, self-reported measure to evaluate symptoms of insomnia, with responses from 0-4 for each question, yielding scores ranging from 0-28. Lower scores represent better outcomes. The primary outcome will be change from enrollment to 8-10 weeks after completion of the intervention.
Time Frame: Collected from the enrollment visit through completion of the primary data collection visit, 8-10 weeks after completion of the intervention
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 56 | 51
units on a scale | -6.98 (0.74) | -4.94 (0.76)

2. Secondary Outcome: Change From Baseline in Sleep Onset Latency and Wake After Sleep Onset
Description: This will be an online daily sleep diary to evaluate the amount and quality of sleep. This allows evaluation of the timing and trajectory of any improvements in sleep, including appreciation of the presence and duration of placebo effects. Measurements of sleep onset latency (SOL) and wake after sleep onset (WASO) were recorded in minutes.
Time Frame: Baseline and 8-10 weeks after completion of intervention
Population: Data was not able to be collected for all participants.
Measure: Mean (Standard Error); unit: minutes
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 47 | 39
minutes
  SOL | -1.00 (0.18) | -0.56 (0.14)
  WASO | -28.42 (8.00) | -22.64 (4.73)

3. Secondary Outcome: Change in Total Sleep Time (TST)
Description: This will be an online daily sleep diary to evaluate the amount and quality of sleep. This allows evaluation of the timing and trajectory of any improvements in sleep, including appreciation of the presence and duration of placebo effects. Participants recorded the total sleep time (TST) they had each night. The outcome indicates the average increase (in hours) of the amount of sleep that each group reported.
Time Frame: as for outcome 1
Population: Data was not able to be collected for all participants.
Measure: Mean (Standard Error); unit: hours
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 47 | 39
hours | 1.15 (0.23) | 0.58 (0.17)

4. Secondary Outcome: Change in RestRefresh and SleepQual
Description: This will be an online daily sleep diary to evaluate the amount and quality of sleep. This allows evaluation of the timing and trajectory of any improvements in sleep, including appreciation of the presence and duration of placebo effects. Participants were asked to report a self-rating on how well they felt rested and refreshed (RestRefresh) and to rate the quality of sleep they had (SleepQual). Both questions were rated on a 0 to 4 scale and higher scores denotes better outcomes for each.
Time Frame: as for outcome 1
Population: Data was not able to be collected for all participants.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 47 | 39
units on a scale
  RestRefresh | 0.60 (0.16) | 0.54 (0.12)
  SleepQual | 0.79 (0.16) | 0.67 (0.12)

5. Secondary Outcome: Change From Baseline in Beck Depression Inventory - II (BDI-II)
Description: Depression will be measured by the Beck Depression Inventory-II (BDI-II). The BDI-II is a 21-item questionnaire with response values of 0-3 for each item, yielding scores ranging from 0-63. Higher scores denotes worse outcomes.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 52 | 49
units on a scale | -3.76 (0.59) | -2.65 (0.61)

6. Secondary Outcome: Change From Baseline in Beck Anxiety Inventory (BAI)
Description: Anxiety will be measured by the Beck Anxiety Inventory (BAI). The BAI is a 21-item questionnaire with response values from 0-3 for each item, yielding scores ranging from 0-63. Higher scores denotes worse outcomes.
Time Frame: as for outcome 1
Population: Data not collected for one participant in the placebo group
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 52 | 48
units on a scale | -0.25 (0.10) | -0.25 (0.10)

7. Secondary Outcome: Change From Baseline in EQ-5D
Description: Health-related quality of life will be measured by the EQ-5D. The EQ-5D consists of 5 items assessing an individual's current health status (values from 0-2), yielding scores ranging from 0-10. Higher scores denotes worse outcomes.
Time Frame: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 52 | 49
units on a scale | 2.73 (1.90) | 0.11 (1.94)

8. Secondary Outcome: Change in Heart Rate Variability (HRV)
Description: Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system (BIOPAC acquisition system and Acknowledge 4.2 software, Santa Barbara, CA), at 1000 Hz, are analyzed using Nevrokard BRS software (Nevrokard BRS, Medistar, Ljubljana, Slovenia). Analysis is conducted on the first complete 5-minute epoch that is considered to be acceptable for analysis. Heart rate variability is measured in the time domain as standard deviation of beat-to-beat interval (SDNN, milliseconds)and the root mean square of successive beat-to-beat differences in R-R interval duration (rMSSD milliseconds). For calculation of SDNN, the R-R intervals are visually inspected, and data considered as artifact is manually removed.
Time Frame: as for outcome 1
Population: Other entries were excluded due to missing or dropped heartbeats and were excluded from the analysis for continuity
Measure: Mean (Standard Error); unit: ms
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 52 | 47
ms
  SDNN | 57.28 (1.34) | 35.81 (1.77)
  rMSSD | 53.06 (5.34) | 26.86 (2.24)

9. Secondary Outcome: Change in Baroflex Sensitivity (BRS)
Description: Blood pressure and heart rate are acquired from 10 minute recordings of noninvasive finger arterial pressure measurements and ECG with participants lying quietly, supine. Systolic BP and beat to beat, RR intervals files generated via the data acquisition system at 1000 Hz, are analyzed using Nevrokard BRS software. Analysis is conducted on the first complete 5-minute epoch. Power spectral densities of systolic blood pressure (SBP) and R-R interval (RRI) oscillations are computed by 512 points Fast Fourier Transform (FFT) and integrated over specified frequency ranges (HF: 0.15-0.4 Hz). The square-root of the ratio of RRI's and SBP powers is computed to calculate HF alpha indices, which reflect BRS. The software scans the RRI and SBP records, identifies sequences, and calculates linear correlation between RRI and SBP for each sequence. The mean of all individual regression coefficients (slopes), a measure of sequence BRS, is then calculated for Sequence UP, DOWN and TOTAL (seq ALL).
Time Frame: 8-10 weeks after completion of the intervention
Population: Other entries were excluded due to missing or dropped heartbeats and were excluded from the analysis for continuity
Measure: Mean (Standard Error); unit: ms/mm Hg
Arm/Group | HIRREM | Placebo
Number analyzed (Participants) | 52 | 47
ms/mm Hg
  HF Alpha | 24.78 (2.17) | 16.26 (1.73)
  Seq ALL | 20.36 (2.03) | 12.31 (1.09)

ADVERSE EVENTS:
Time Frame: 16-18 weeks after completion of the intervention
Arm/Group | HIRREM | Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/51
Other Adverse Events (participants affected / at risk) | 6/56 | 7/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIRREM (N=56) | Placebo (N=51)
Change in sleep (General disorders) | 2 | 2 — Change in sleep beyond baseline threshold
Change in emotions or awareness of feelings (Social circumstances) | 1 | 2
Head fullness (General disorders) | 3 | 2 — Mild headache
Skin irritation at scalp sensor site (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes